CLINICAL TRIAL: NCT04762186
Title: A Phase I/ Randomized Phase II Trial to Analyse Safety and Efficacy of Human SARS-CoV-2-specific T Lymphocyte Transfer in Patients With COVID-19 in Need of Treatment or at Risk of Severe COVID-19
Brief Title: Viable Human SARS-CoV-2 Specific T Cell Transfer in Patients at Risk for Severe COVID-19
Acronym: ACT-COVID-19
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Universitätsklinikum Köln (Other)
Collaborators: ZKS Köln (Other); Hannover Medical School (Other); Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-4480
Record Dates: First submitted 2021-02-11; First posted 2021-02-21 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Moderate COVID-19-infection
Keywords: COVID-19; T-Cell; SARS-CoV-2; Infusion; Adoptive; Allogeneic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This trial consist of an open-label dose escalation phase in SARS-CoV-2 infected participants.
Masking Description: During the dose-escalation phase, the study participants and the study team are aware of the treatment as this is an open label trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation (Experimental): SARS CoV-2 infected participants will receive a single infusion over 15 to 30 minutes
  Interventions: Drug: human SARS-CoV 2 specific T lymphocytes

INTERVENTIONS:
Drug: human SARS-CoV 2 specific T lymphocytes — In dose level one, SARS-CoV-2 infected patients will receive 1,000 viable human SARS CoV-2 specific T lymphocytes per kg BW.
  In dose level two SARS-CoV-2 infected patients will receive 5,000 viable human SARS CoV-2 specific T lymphocytes per kg BW.
  In parallel, all patients will receive the current SoC treatment for COVID-19.

SUMMARY:
Monocentric open phase I (dose escalation component), followed by a multi-center, randomized, phase II component benchmarking IMP+SoC against SoC

DETAILED DESCRIPTION:
The clinical trial will consist of a phase I and a phase II part. The main trial objective in the phase I part is to determine the recommended phase II dose (RP2D) of viable human SARS-CoV 2-specific T cells by evaluation of safety and tolerability.

In the phase II part, the primary objective is to gain first data on efficacy of adaptive therapy with viable human SARS-CoV-2-specific T cells. This will be a randomized, prospective feasibility trial.

Details to phase II will be updated after completion of phase I.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above
* Written informed consent from the trial subject has been obtained
* Willing to follow contraception guidelines
* Tested positive for SARS-CoV-2 by PCR <72 hours after swab
* A maximum of 14 days between onset of symptoms and enrollment
* WHO score 5 OR
* WHO score 4 with at least one additional risk factor for disease progression
* Acceptable risk factors are:

  * Radiographically proven lung infiltrates
  * Immunosuppression either by malignant disease or it's treatment, or other underlying diseases leading to immunodeficiency or underlying diseases that require treatment resulting in immunosuppression
  * Immunosuppressive drugs or steroids at a prednisolone equivalent of <1 mg/kg BW)
  * Receipt of an autologous transplant within the last 5 years
  * Receipt of an allogeneic transplant within the last 5 years or ongoing immunosuppression

Exclusion criteria:

* Participation in any other clinical trial of an experimental agent treatment
* Active GvHD or history of GvHD
* History of CAR-T-Cell Therapy
* COVID-19 WHO ordinal scale ≥6
* Anticipated life-expectancy <72 hours
* Expected duration of hospital stay <72 hours
* Sepsis-induced leukopenia or thrombocytopenia (leukocytes <1,000/µl or platelets <50,000/µl). If the cytopenias result from underlying hematologic disease or its treatment this will not be regarded as exclusion criterion
* CT pneumonia score ≥13 [50]
* Any Steroids ≥1 mg/kg Prednisolon-equivalent/kg BW, besides 6 mg Dexamethasone i.v. or p.o. 1x/d as SoC for COVID-19
* Pregnant or breast feeding
* Any serious medical condition or abnormality of clinical laboratory tests that, in the Investigator's judgment, precludes the subject's safe participation in and completion of the study
* Therapeutic donor lymphocyte infusion (DLI) less than 100 days prior to IMP infusion
* Known hypersensitivity to iron dextran
* Known pre-existing human anti-mouse antibodies (HAMAs)
* ontraindication against mandatory protocol-inherent comedication(s): antihistamine and/or acetaminophen
* Failure to use highly-effective contraceptive methods. The following contraceptive methods with a Pearl Index lower than 1% are regarded as highly-effective:

  * Oral hormonal contraception ('pill')
  * Dermal hormonal contraception
  * Vaginal hormonal contraception (NuvaRing®)
  * Contraceptive plaster
  * Long-acting injectable contraceptives
  * Implants that release progesterone (Implanon®)
  * Tubal ligation (female sterilization)
  * Intrauterine devices that release hormones (hormone spiral)
  * Double barrier methods
  * This means that the following are not regarded as safe: condom plus spermicide, simple barrier methods (vaginal pessaries, condom, female condoms), copper spirals, the rhythm method, basal temperature method, and the withdrawal method (coitus interruptus).
* Persons with any kind of dependency on the principal investigator or employed by the sponsor or principal investigator
* Legally incapacitated persons
* Persons held in an institution by legal or official order

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Phase I: Dose-limiting toxicities | 28 days
  Dose-limiting toxicities until Day 28 after infusion of SARS-CoV-2- specific T cells

SECONDARY OUTCOMES:
Phase I: Safety | 3 Month
  The rate and severity of adverse events after infusion of SARS-CoV-2 specific T cells during the trial
Phase I: Acute graft- vs. -host disease | 100 days after enrollment
  Clinical manifestations of acute graft- vs. -host disease at day 100 after randomization
Phase I: Clinical status | 100 days after enrollment
  Clinical status as assessed on the WHO ordinal scale
Phase I: Hospitalization | 100 days after enrollment
  duration in days
Phase I: SARS-CoV-2 PCR positivity | 100 days after enrollment
  Duration of SARS-CoV-2 PCR positivity (in days) from nasooropharyngeal swabs until discharge or death
Phase I: Detection of viable human SARS-CoV-2-specific T lymphocyte | 100 days after enrollment
  Detection of viable human SARS-CoV-2-specific T lymphocyte after infusion
Phase I: viral shedding in nasooropharyngeal swabs | 100 days after enrollment
  Effect of viable human SARS-CoV-2-specific T lymphocyte infusion on viral shedding in nasooropharyngeal swabs

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Köhler, Dr., Principal Investigator — Department I for Internal Medicine University Hospital of Cologne
Locations (1):
- Department I for Internal Medicine University Hospital of Cologne, Cologne, North Rhine-Westphalia, Germany